CLINICAL TRIAL: NCT01464983
Title: A Multicentre Randomised Parallel-groups Double-blind Double-dummy Single-dose Study to Compare Acetylsalicylic Acid 500 mg and 1,000 mg With Ibuprofen 200 mg and 400 mg and Placebo for Tolerability and Efficacy in the Treatment of Episodic Tension-type Headache
Brief Title: Placebo and Active Controlled, Double Dummy Study to Compare Efficacy of Aspirin and Ibuprofen in Treatment of Episodic Tension-type Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11220
Record Dates: First submitted 2011-05-17; First posted 2011-11-04 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Headache; Tension-Type Headache; Tension-Type Headache (Episodic)
MeSH Terms: conditions — Headache; Tension-Type Headache; Recurrence | interventions — Aspirin; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)
- Arm 2 (Experimental)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)
- Arm 3 (Active Comparator)
  Interventions: Drug: Ibuprofen
- Arm 4 (Active Comparator)
  Interventions: Drug: Ibuprofen
- Arm 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) — Acetylsalicylic acid 500 mg orally, single dose, 1 tablet; in addition, 1 Placebo tablet of Acetylsalicylic acid, and 2 Placebo tablets of Ibuprofen
  Arms: Arm 1
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) — Acetylsalicylic acid 2 x 500 mg orally, single dose, 2 tablets; in addition, 2 Placebo tablets of Ibuprofen
  Arms: Arm 2
Drug: Ibuprofen — Ibuprofen 200 mg orally, single dose, 1 tablet; in addition, 1 Placebo tablet of Ibuprofen, and 2 Placebo tablets of Acetylsalicylic Acid
  Arms: Arm 3
Drug: Ibuprofen — Ibuprofen 2 x 200 mg orally, single dose, 2 tablets; in addition, 2 Placebo tablets of Acetylsalicylic Acid
  Arms: Arm 4
Drug: Placebo — 2 Placebo tablets of Acetylsalicylic Acid, and 2 Placebo tablets of Ibuprofen, orally, single dose
  Arms: Arm 5

SUMMARY:
The purpose of this study is to determine the efficacy and tolerability of 500 mg and 1000 mg Aspirin® (study medication) by comparing it to placebo (the control group without active substance) or 200 mg or 400 mg Ibuprofen (study medication) in treating the symptoms of episodic tension-type headache. The study is designed to develop a treatment method against episodic tension-type headache which will have more advantages for patients than the methods that are currently available.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female, 18 to 65 years of age
* Normal blood pressure
* Patients suffering from episodic tension-type headache
* Headache lasting from 30 minutes to 7 days
* Headache had at least two of the following characteristics:

Bilateral location. Pressing/tightening (non-pulsating). Mild or moderate intensity. Not aggravated by routine physical activity such as walking or climbing stairs.

- Both of the following: No nausea or vomiting. No more than one of photophobia or phonophobia.

Exclusion Criteria:

* Other headaches, including migraine, that required medical treatment
* Hypersensitivity to acetylsalicylic acid, salicylates, ibuprofen or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Serious physical illness especially uncontrolled disorders of kidney, liver, lung, heart or brain function, neurological disorders or severe chronic or terminal disease
* Mental illness, including depression
* Needed or were using or likely to need or use any of the prohibited concomitant medications: antidepressants, oxicams
* Pregnant or lactating women, or sexually active women of child-bearing potential unless using effective contraception
* Participating in any other clinical study or had done within the previous 4 weeks
* Had been previously enrolled in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1115 (Actual)
Dates: Start 2004-01; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with total or meaningful headache relief at 2 hours after intake of study medication | 2 hours post dose

SECONDARY OUTCOMES:
Headache pain relief measured serially on a categorical scale | Until 4 hours post dose
Measuring the functional ability on conducting everydays activity on a 4 point categorical scale | 2 and 24 hours post dose
Global assessment of pain therapy | 24 hours post dose
Safety - assessment of adverse events | Up to 10 weeks after screening

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- United Kingdom (10):
  - Reading, Berkshire
  - Manchester, Greater Manchester
  - Chorley, Lancashire
  - Wigan, Lancashire
  - Liverpool, Merseyside
  - Cardiff, South Glamorgan
  - Glasgow, Strathclyde
  - Birmingham, West Midlands
  - Coventry, West Midlands
  - Wolverhampton, West Midlands